CLINICAL TRIAL: NCT05678634
Title: Optimizing Feedback-based Learning in Children With Developmental Language Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MGH Institute of Health Professions (Other)
Responsible Party: Principal Investigator, Yael Arbel, Professor, MGH Institute of Health Professions
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022P003376
Record Dates: First submitted 2023-01-03; First posted 2023-01-10 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Developmental Language Disorder
MeSH Terms: conditions — Language Development Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Children with developmental language disorder (Experimental)
  Interventions: Behavioral: Declarative learning with immediate feedback; Behavioral: Declarative learning with delayed feedback; Behavioral: Probabilistic learning with immediate feedback; Behavioral: Probabilistic learning with delayed feedback; Behavioral: Word learning task with active feedback; Behavioral: Word learning task with passive feedback

INTERVENTIONS:
Behavioral: Declarative learning with immediate feedback — Children will complete a paired associate learning task on a computer. Each response on half of the blocks will be followed by performance feedback. Feedback will be provided 500 ms following a response (button press)
Behavioral: Declarative learning with delayed feedback — Children will complete a paired associate learning task on a computer. Each response on half of the blocks will be followed by performance feedback. Feedback will be provided 5000 ms following a response (button press)
Behavioral: Probabilistic learning with immediate feedback — Children will complete a probabilistic learning task on a computer. Each response on half of the blocks will be followed by feedback. Feedback will be provided 500 ms following a response (button press)
Behavioral: Probabilistic learning with delayed feedback — Children will complete a probabilistic learning task on a computer. Each response on half of the blocks will be followed by feedback. Feedback will be provided 5000 ms following a response (button press)
Behavioral: Word learning task with active feedback — Children will complete a two-choice nonword learning task in which they will be tasked with learning to associate novel objects with novel nonword names through trial and error guided by feedback. Each response will be followed by feedback either indicating that the response is correct or prompting the child to try again (i.e., to correct an error)
Behavioral: Word learning task with passive feedback — Children will complete a two-choice nonword learning task in which they will be tasked with learning to associate novel objects with novel nonword names. Regardless of response accuracy on each trial, each response will be followed by a visual presentation of the correct response.

SUMMARY:
This project aims to optimize a critical but understudied ingredient of language intervention provided to children with developmental language disorder (DLD) - feedback. The project will bridge a gap between previous findings in our lab of inefficient feedback processing in DLD and clinical practice by identifying the conditions under which feedback-based learning can be improved in DLD. The investigators hypothesize that the effectiveness of feedback can be significantly enhanced for children with DLD when it is tailored to their unique learning strengths. The rationale for this project is based on evidence that feedback-based learning can be improved by enhancing the dominance of an intact learning system. The project will achieve its aim by manipulating (1) the timing of the feedback (immediate vs. delayed) and (2) the level of the learner's involvement in error correction dictated by feedback (active vs. passive correction). Aim 1 will determine the effect of manipulating feedback timing on learning in 140 school-age children (8-12 years) with DLD. While immediate feedback is processed by the striatum, which is also implicated in implicit learning, delaying the feedback by a few seconds shifts feedback processing to the mediate temporal lobe (MTL)-based declarative learning system. Evidence that delaying feedback improves learning in DLD would support the hypothesis of the implicit deficit theory that intervention should capitalize on declarative learning mechanisms. The project will test a novel alternative feedback-learning parity hypothesis whereby feedback-based learning is optimized when the timing of the feedback is aligned with the dominant learning system at a given time (i.e., immediate feedback during striatal-based probabilistic learning; delayed feedback during MTL-based declarative learning). Within the same group of children, Aim 2 will compare feedback-based learning in children with DLD when feedback (a) prompts active self-correction or (b) passively exposes learners to error corrections (corrective recast). Children will engage in two nonword-object paired-associate learning tasks. In one task, feedback will promote active self-correction, which is in line with declarative learning. In the other task, feedback will passively expose the learner to corrective feedback in a manner consistent with teaching approaches aiming at reducing awareness of errors. The project will determine whether children with DLD learn better when feedback prompts self-correction or when they are exposed to passive corrections. Electrophysiological measures will indicate whether passive corrections (corrective recast) are processed as negative feedback by children with DLD. For both aims, behavioral indicators of response to feedback will be complemented by electrophysiological measures of feedback processing that can determine the involvement of the striatum and MTL brain systems during the learning process. This work is scientifically and clinically significant because elucidating what manipulations optimize feedback-based learning will enhance our understanding of the impaired learning mechanism in DLD and will provide clinical guidance on what type of feedback to use during an intervention.

ELIGIBILITY:
Inclusion Criteria:

* English as the primary language Nonverbal intelligence quotient (IQ) score on the Wechsler Intelligence Scale for Children-5th Edition (WISC-V) Standard Score >70 Identification Core score on the Test of Integrated Language & Literacy Skills (TILLS) equal to or less than 34

Exclusion Criteria:

* Hearing loss or other known neurological deficits, or diagnoses (e.g., Autism, Traumatic Brain Injury)
* Evidence of color blindness as measured by the EnChroma computer base color blindness screening test for children

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy (percent correct) on a two-choice paired associate test immediately after the task | Immediately after learning task
  Accuracy on a two-choice paired-associate test following each of the learning conditions. The structure of a test trial will be similar to the structure of a task trial but it will not include feedback. This measure will evaluate learning outcomes.
Accuracy (percent correct) on a two-choice paired associate test 1 week after the task | 1 week after the learning task
  Accuracy on a two-choice paired-associate test a week after the completion of each learning task. The structure of a test trial will be similar to the structure of a task trial but it will not include feedback. This measure will evaluate learning retention.
FRN amplitude | During each learning task
  The amplitude (in microvolts) of the feedback related negativity (FRN) event related potential
N170 amplitude | During each learning task
  The amplitude (in microvolts) of the N170 event related potential

CONTACTS AND LOCATIONS:
Overall Officials: Yael Arbel, PhD, Principal Investigator — MGH Institute of Health Professions
Locations (1):
- MGH Institute of Health Professions, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No